CLINICAL TRIAL: NCT04060680
Title: Extravascular ICD Pivotal Study (EV ICD)
Brief Title: Extravascular ICD Pivotal Study
Acronym: EV ICD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: U1111-1236-4810; MDT16028 (Other: Medtronic)
Record Dates: First submitted 2019-08-14; First posted 2019-08-19 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-04

CONDITIONS: Tachycardia; Ventricular Arrythmia
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Implant Attempt (Experimental): Patients will be implanted with an extravascular ICD and undergo requisite electrical testing.
  Interventions: Device: Defibrillation using the Extravascular ICD
- Continued Access Implant Attempt (Experimental): Continued Access for United States
  Interventions: Device: Defibrillation using the Extravascular ICD

INTERVENTIONS:
Device: Defibrillation using the Extravascular ICD — VT/VF induction attempted for defibrillation testing, as well as requisite electrical testing.

SUMMARY:
Pivotal Summary:

The study is designed to demonstrate safety and efficacy of the Extravascular Implantable Cardioverter Defibrillator (EV ICD) System.

Continued Access Summary:

This study is designed to provide continued access to the Extravascular Implantable Cardioverter Defibrillator (EV ICD) System.

DETAILED DESCRIPTION:
The study will enroll subjects who are indicated to receive an implantable defibrillator and who meet all of the inclusion criteria and none of the exclusion criteria. Subjects will receive an investigational Extravascular Implantable Cardioverter Defibrillator (EV ICD) system, in which a lead is placed outside of the heart and veins to deliver defibrillation therapy. Subjects will be followed until regulatory approval is received.

ELIGIBILITY:
Pivotal Inclusion Criteria:

* Patient has a Class I or IIa indication for implantation of an ICD according to the ACC/AHA/HRS Guidelines [i], or ESC guidelines [ii].
* Patient is at least 18 years of age and meets age requirements per local law.
* Patient is geographically stable and willing and able to complete the study procedures and visits for the duration of the follow-up.

  [i] Al-Khatib SM, Stevenson WG, Ackerman MJ, Bryant WJ, Callans DJ, Curtis AB, Deal BJ, Dickfeld T, Field ME, Fonarow GC, Gillis AM, Hlatky MA, Granger CB, Hammill SC, Joglar JA, Kay GN, Matlock DD, Myerburg RJ, Page RL. 2017 AHA/ACC/HRS guideline for management of patients with ventricular arrhythmias. [ii] Priori SG, Blomstrom-Lundqvist C, Mazzanti A, Blom N, Borggrefe M, Camm J, Elliot PM, Fitzsimons D, Hatala R, Hindricks G, Kirchhof P, Kjeldsen K, Kuck KH, Hernandez-Madrid A, Nikolaou N, Norekval TM, Spaulding C, Van Veldhuisen DJ. 2015 ESC guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death. European Heart Journal 2015 36:41 (2793-2867). https://doi.org/10.1093/eurheartj/ehv316

Pivotal Exclusion Criteria:

* Patient is unwilling or unable to personally provide Informed Consent.
* Patient has indications for bradycardia pacing [iii] or Cardiac Resynchronization Therapy (CRT) [iv] (Class I, IIa, or IIb indication).
* Patient with an existing pacemaker, ICD, or CRT device implant or leads.
* Patients with these medical interventions are excluded from participation in the study:

  * Prior sternotomy
  * Any prior medical condition or procedure that leads to adhesions in the anterior mediastinal space (i.e., prior mediastinal instrumentation, mediastinitis)
  * Prior abdominal surgery in the epigastric region
  * Planned sternotomy
  * Prior chest radiotherapy

Or any other prior/planned medical intervention not listed that precludes their participation in the opinion of the Investigator.

* Patient has previous pericarditis that:

  * Was chronic and recurrent, or
  * Resulted in pericardial effusion [v], or
  * Resulted in pericardial thickening or calcification [vi].
* Patients with these medical conditions or anatomies are excluded from participation in the study:

  * Hiatal hernia that distorts mediastinal anatomy
  * Marked sternal abnormality (e.g., pectus excavatum)
  * Decompensated heart failure
  * COPD with oxygen dependence
  * Gross hepatosplenomegaly

Or any other known medical condition or anatomy type not listed that precludes their participation in the opinion of the Investigator.

* Patients with a medical condition that precludes them from undergoing defibrillation testing:

  * Severe aortic stenosis
  * Intracardiac LA or LV thrombus
  * Severe proximal three-vessel or left main coronary artery disease without revascularization
  * Hemodynamic instability
  * Unstable angina
  * Recent stroke or transient ischemic attack (within the last 6 months)
  * Known inadequate external defibrillation
  * LVEF <20%
  * LVEDD >70 mm

Or any other known medical condition not listed that precludes their participation in the opinion of the Investigator.

* Patient with any evidence of active infection or undergoing treatment for an infection.
* Patient is contraindicated from temporary suspension of oral/systemic anticoagulation
* Patient with current implantation of neurostimulator or any other chronically implanted device that delivers current in the body.
* Patient meets ACC/AHA/HRS or ESC clinical guideline Class III criteria for an ICD (e.g., life expectancy of less than 12 months).
* Patient is enrolled or planning to enroll in a concurrent clinical study that may confound the results of this study, without documented pre-approval from a Medtronic study manager.
* Patient with any exclusion criteria as required by local law (e.g., age or other).
* Pregnant women or breastfeeding women, or women of child bearing potential and who are not on a reliable form of birth regulation method or abstinence.

[iii] 2015 HRS/EHRA/APHRS/SOLAECE expert consensus statement on optimal implantable cardioverter-defibrillator programming and testing). [iv] ACC/AHA/HRS guidelines for Cardiac Resynchronization Therapy. [v] As documented on echo or MRI. [vi] As documented on CT scan or MRI.

Continued Access Inclusion Criteria

1. Patient has a Class I or IIa indication for implantation of an ICD according to the ACC/AHA/HRS Guidelines.[1]
2. Patient is willing and able to sign and date the Informed Consent Form for their participation in the study.
3. Patient is at least 18 years of age and meets age requirements per local law.
4. Patient is geographically stable and willing and able to comply with the study procedures and visits for the duration of the follow-up.

[1] Al-Khatib SM, Stevenson WG, Ackerman MJ, Bryant WJ, Callans DJ, Curtis AB, Deal BJ, Dickfeld T, Field ME, Fonarow GC, Gillis AM, Granger CB, Hammill SC, Hlatky MA, Joglar JA, Kay GN, Matlock DD, Myerburg RJ, Page RL. 2017 AHA/ACC/HRS Guideline for Management of Patients With Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2018 Oct 2;72(14):e91-e220. doi: 10.1016/j.jacc.2017.10.054. Epub 2018 Aug 16. Review. Erratum in: J Am Coll Cardiol. 2018 Oct 2;72(14):1760.

Continued Access Exclusion Criteria

1. Patient has indications for bradycardia pacing[2] or Cardiac Resynchronization Therapy (CRT)[3] (Class I, IIa, or IIb indication).
2. Patients with an existing pacemaker, ICD, or CRT device or leads.
3. Patients with these medical interventions are excluded from participation in the study:

   * Prior sternotomy
   * Any prior medical condition or procedure that leads to adhesions in the anterior mediastinal space (i.e., prior mediastinal instrumentation, mediastinitis)
   * Prior abdominal surgery in the epigastric region
   * Planned sternotomy
   * Prior chest radiotherapy Or any other prior/planned medical intervention not listed that precludes their participation in the opinion of the Investigator.
4. Patients with these medical conditions or anatomies are excluded from participation in the study:

   * Hiatal hernia that distorts mediastinal anatomy
   * Marked sternal abnormality (e.g., pectus excavatum that impedes the substernal tunneling path or procedure)
   * Decompensated heart failure
   * COPD with oxygen dependence
   * Gross hepatosplenomegaly Or any other known medical condition or anatomy type not listed that precludes their participation in the opinion of the Investigator.
5. Patients with a medical condition that precludes them from undergoing defibrillation testing:

   * Severe aortic stenosis
   * Current Intracardiac LA or LV thrombus
   * Severe proximal three-vessel or left main coronary artery disease without revascularization
   * Hemodynamic instability
   * Unstable angina
   * Recent stroke or transient ischemic attack (within the last 6 months)
   * Known inadequate external defibrillation
   * LVEF < 20%
   * LVEDD >70 mm Or any other known medical condition not listed that precludes their participation in the opinion of the Investigator.
6. Patient with any evidence of active infection or undergoing treatment for an infection.
7. Patient is contraindicated from temporary suspension of oral/systemic anticoagulation.
8. Patient with current implantation of neurostimulator or any other chronically implanted device that delivers current in the body.
9. Patient meets ACC/AHA/HRS or ESC clinical guideline Class III criteria for an ICD (e.g., life expectancy of less than 12 months).
10. Patient is enrolled or planning to enroll in a concurrent clinical study that may confound the results of this study, without documented pre-approval from a Medtronic study manager.
11. Patient with any exclusion criteria as required by local law (e.g., age or other).
12. Pregnant women or breastfeeding women, or women of childbearing potential and who are not on a reliable form of birth regulation method or abstinence* (*If required by local law, women of child-bearing potential must undergo a pregnancy test within seven days prior to EV ICD Continued Access Study procedures)

[2] Wilkoff BL, Fauchier L, Stiles MK, Morillo CA, Al-Khatib SM, Almendral J, Aguinaga L, Berger RD, Cuesta A, Daubert JP, Dubner S, Ellenbogen KA, Mark Estes NA 3rd, Fenelon G, Garcia FC, Gasparini M, Haines DE, Healey JS, Hurtwitz JL, Keegan R, Kolb C, Kuck KH, Marinskis G, Martinelli M, McGuire M, Molina LG, Okumura K, Proclemer A, Russo AM, Singh JP, Swerdlow CD, Teo WS, Uribe W, Viskin S, Wang CC, Zhang S. 2015 HRS/EHRA/APHRS/SOLAECE expert consensus statement on optimal implantable cardioverter-defibrillator programming and testing. Heart Rhythm. 2016 Feb;13(2):e50-86.

doi: 10.1016/j.hrthm.2015.11.018. Epub 2015 Dec 1. [3] Kusumoto FM, Schoenfeld MH, Barrett C, Edgerton JR, Ellenbogen KA, Gold MR, Goldschlager NF, Hamilton RM, Joglar JA, Kim RJ, Lee R, Marine JE, McLeod CJ, Oken KR, Patton KK, Pellegrini CN, Selzman KA, Thompson A, Varosy PD. 2018 ACC/AHA/HRS Guideline on the Evaluation and Management of Patients With Bradycardia and Cardiac Conduction Delay: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2019 Aug 20;74(7):e51-e156. doi: 10.1016/j.jacc.2018.10.044. Epub 2018 Nov 6. Erratum in: J Am Coll Cardiol. 2019 Aug 20;74(7):1016-1018.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2024-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Friedman, MD, Principal Investigator — Mayo Clinic
Locations (56):
- United States (33):
  - HonorHealth Cardiac Arrhythmia Group - Osborn, Scottsdale, Arizona
  - University of California San Diego (UCSD), La Jolla, California
  - Continued Access: Sequoia Hospital, Redwood City, California
  - Sequoia Hospital, Redwood City, California
  - Continued Access: Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - MedStar Wahsington Hospital Center, Washington D.C., District of Columbia
  - Baptist Health, Jacksonville, Florida
  - Continued Access: Baptist Health, Jacksonville, Florida
  - AdventHealth Cardiovascular Research Institute, Orlando, Florida
  - Northwestern University, Chicago, Illinois
  - Prairie Education & Research Cooperative, Springfield, Illinois
  - Iowa Heart Center, Des Moines, Iowa
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Continued Access: University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Continued Access: Saint Luke's Mid America Heart Institute, Kansas City, Missouri
  - Saint Luke's Mid America Heart Institute, Kansas City, Missouri
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Continued Access: Lourdes Cardiology Services, Voorhees Township, New Jersey
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - Continued Access: North Shore University Hospital, Manhasset, New York
  - North Shore Uniersity Hospital, Manhasset, New York
  - New York-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - Continued Access: New York-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - Duke University Medical Center (DUMC), Durham, North Carolina
  - Continued Access: University Hospitals Cleveland Clinic Medical Center, Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Continued Access: OhioHealth Research and Innovation Institute (OHRI), Columbus, Ohio
  - OhioHealth Research and Innovation Institute (OHRI), Columbus, Ohio
  - University of Washington (UW) Medical Center, Seattle, Washington
- Australia (4):
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre Clayton, Clayton, Victoria
  - Austin Hospital, Heidelberg, Victoria
- Kepler Universitätsklinikum Med Campus III., Linz, Austria
- Canada (2):
  - London Health Sciences Centre - University Campus, London
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ), Québec
- Odense Universitetshospital, Odense, Denmark
- France (2):
  - CHRU de Tours - Hôpital Trousseau, Chambray-lès-Tours
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Semmelweis Egyetem AOK, Budapest, Hungary
- Policlinico Sant' Orsola - Malpighi, Bologna, Italy
- Netherlands (3):
  - Amsterdam UMC - Locatie AMC, Amsterdam
  - St. Antonius Ziekenhuis, Nieuwegein
  - Isala Zwolle, Zwolle
- Christchurch Hospital, Christchurch, New Zealand
- Oslo Universitetssykehus-Rikshospitalet, Oslo, Norway
- Narodowy Instytut Kardiologii - Stefana kardynała Wyszyńskiego, Warsaw, Poland
- The College of Medicine & King Khalid University Hospital, King Saud University, Riyadh, Saudi Arabia
- Hospital Universitario Reina Sofía, Córdoba, Spain
- UniversitätsSpital Zürich, Zurich, Switzerland
- King's College of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Friedman P, Murgatroyd F, Boersma LVA, Manlucu J, Knight BP, Clementy N, Leclercq C, Amin A, Merkely B, Birgersdotter-Green UM, Chan JYS, Biffi M, Knops RE, Engel G, Munoz Carvajal I, Epstein LM, Sagi V, Johansen JB, Sterlinski M, Steinwender C, Hounshell T, Abben R, Thompson AE, Zhang Y, Wiggenhorn C, Willey S, Crozier I; Extravascular ICD Pivotal Study Investigators. Performance and Safety of the Extravascular Implantable Cardioverter Defibrillator Through Long-Term Follow-Up: Final Results From the Pivotal Study. Circulation. 2025 Jan 28;151(4):322-332. doi: 10.1161/CIRCULATIONAHA.124.071795. Epub 2024 Sep 26. PMID 39327797
- [Derived] Swerdlow C, Gillberg J, Boersma LVA, Manlucu J, Zhang X, Zhang Y, Hernandez AA, Bhatia V, Murgatroyd F. Extravascular Implantable Cardioverter-Defibrillator Sensing and Detection in a Large Global Population. JACC Clin Electrophysiol. 2024 Aug;10(8):1896-1912. doi: 10.1016/j.jacep.2024.02.033. Epub 2024 May 15. PMID 38752961
- [Derived] Friedman P, Murgatroyd F, Boersma LVA, Manlucu J, O'Donnell D, Knight BP, Clementy N, Leclercq C, Amin A, Merkely BP, Birgersdotter-Green UM, Chan JYS, Biffi M, Knops RE, Engel G, Munoz Carvajal I, Epstein LM, Sagi V, Johansen JB, Sterlinski M, Steinwender C, Hounshell T, Abben R, Thompson AE, Wiggenhorn C, Willey S, Crozier I; Extravascular ICD Pivotal Study Investigators. Efficacy and Safety of an Extravascular Implantable Cardioverter-Defibrillator. N Engl J Med. 2022 Oct 6;387(14):1292-1302. doi: 10.1056/NEJMoa2206485. Epub 2022 Aug 28. PMID 36036522
- [Derived] Crozier I, O'Donnell D, Boersma L, Murgatroyd F, Manlucu J, Knight BP, Birgersdotter-Green UM, Leclercq C, Thompson A, Sawchuk R, Willey S, Wiggenhorn C, Friedman P. The extravascular implantable cardioverter-defibrillator: The pivotal study plan. J Cardiovasc Electrophysiol. 2021 Sep;32(9):2371-2378. doi: 10.1111/jce.15190. Epub 2021 Aug 5. PMID 34322918

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first site was activated on 13SEP2019. The first EV ICD Pivotal subject was enrolled on 16SEP2019 and implanted on the same day. The last subject enrollment occurred on 14OCT2021, and the last implant occurred on 15OCT2021. Sites were notified of enrollment completion on 18OCT2021.
Pre-assignment Details: Among 356 enrolled subjects, 40 exited the study without having an implant attempt of the Extravascular ICD System due to: adverse event (2), physician decision (7), procedure not attempted (4), sponsor request (1), withdrawal by subject (10), and other reasons (16).
Groups:
- Implant Attempt: Subjects undergoing an implant attempt of an Extravascular ICD System, including implant testing (sensing, impedance and pacing testing) and induction and defibrillation testing using the Extravascular ICD.
- Continued Access Implant Attempt: Continued Access
Period: Overall Study
Arm/Group | Implant Attempt | Continued Access Implant Attempt
Started | 316 (Subjects who underwent an implant attempt of the Extravascular ICD System) | 33
Completed | 292 (Subjects followed up at least to the 6-month visit after the Extravascular ICD System having been fully implanted) | 31
Not Completed | 24 | 2
Not completed — Unsuccessful implant | 17 | 2
Not completed — Adverse Event | 3 | 0
Not completed — Death | 2 | 0
Not completed — Study product no longer in use | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who underwent an implant attempt of the Extravascular ICD System
Groups:
- Implant Attempt Pivotal; Implant Attempt Continued Access: Subjects undergoing an implant attempt of an Extravascular ICD System, including implant testing (sensing, impedance and pacing testing) and induction and defibrillation testing using the Extravascular ICD.
- Total: Total of all reporting groups
Arm/Group | Implant Attempt Pivotal | Implant Attempt Continued Access | Total
Number analyzed (Participants) | 316 | 33 | 349
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (13.1) | 49.2 (13.9) | 53.4 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 9 | 89
  Male | 236 | 24 | 260
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 9
  Not Hispanic or Latino | 110 | 29 | 139
  Unknown or Not Reported | 199 | 2 | 201
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 7 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 16 | 8 | 24
  White | 87 | 21 | 108
  More than one race | 6 | 0 | 6
  Unknown or Not Reported | 197 | 2 | 199
New York Heart Association [Count of Participants; unit: Participants]
  Class I: No symptoms and no limitations in ordinary physical activity. | 75 | 4 | 79
  Class II: Slight limitation of physical activity. | 184 | 15 | 199
  Class III: Marked limitation of physical activity. | 23 | 3 | 26
  Class IV: Unable to carry on any physical activity without discomfort. Symptoms at rest. | 0 | 0 | 0
  Classification Not Available | 34 | 1 | 35
  No Heart Failure | 0 | 10 | 10
ICD Indication [Count of Participants; unit: Participants]
  Primary Prevention | 258 | 17 | 275
  Secondary Prevention | 57 | 15 | 72
  Other | 1 | 1 | 2
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.0 (5.6) | 31 (8) | 28.3 (5.9)
Region [Count of Participants; unit: Participants]
  Asia Pacific | 37 | 0 | 37
  Europe, Middle East, and Africa | 159 | 0 | 159
  North America | 120 | 33 | 153

OUTCOME MEASURES:

1. Primary Outcome: Safety Outcome - Freedom From Major Complications Related to the EV ICD System and/or Procedure at 6 Months Post-implant
Description: The primary safety endpoint is defined as a subject's first occurrence of a major complication related to the EV ICD System and/or procedure, as determined by an independent Clinical Events Committee (CEC), that occurs on or prior to 6 months (182 days) post-implant.
Time Frame: 6 Months (182 days) post implant
Population: Subjects who underwent an implant attempt of the Extravascular ICD System
Measure: Count of Participants; unit: Participants
Arm/Group | Implant Attempt
Number analyzed (Participants) | 316
Participants | 293
Statistical Analysis 1: Comparison: Implant Attempt; The primary safety objective is to demonstrate the freedom from major complications related to the EV ICD System and/or procedure at 6 months post-implant exceeds an OPC of 79%. H0: p ≤ 0.79 HA: p > 0.79, where p denotes the 6-month (182 days) freedom from major EV ICD System/procedure-related complications rate; Test type: Superiority — The pre-specified Objective Performance Criterion (OPC) for the major complication free rate at 6 months is 0.79. If the lower confidence bound of two-sided 95% confidence interval for the freedom from the first major EV ICD System/procedure-related complication through 182 days post implant exceeds 0.79, the primary safety objective will be met. The freedom from the first major EV ICD System/procedure-related complication was estimated using the Kaplan-Meier method; p < 0.0001, Kaplan-Meier method — A priori threshold for statistical significance is 0.025; Major complication-free rate = 92.6, 95% CI 2-sided [89.0 to 95.0]

2. Primary Outcome: Efficacy Outcome - Defibrillation Efficacy at Implant of the EV ICD System
Description: Each subject will demonstrate a successful defibrillation outcome if either 2 successive induced ventricular fibrillation episodes are terminated by the subject's device delivering a shock at the required energy level, or if one such episode is successfully terminated by the subject's device delivering a shock at a lower energy level. Up to 6 such episodes may be induced to test device efficacy.
Time Frame: At Implant
Population: Subjects who completed the implant defibrillation testing protocol
Measure: Count of Participants; unit: Participants
Groups:
- Implant Defibrillation Testing: Subjects undergoing an implant attempt of an Extravascular ICD System, including implant testing (sensing, impedance and pacing testing) and induction and defibrillation testing using the Extravascular ICD.
Arm/Group | Implant Defibrillation Testing
Number analyzed (Participants) | 302
Participants | 298
Statistical Analysis 1: Comparison: Implant Defibrillation Testing; The primary efficacy is to demonstrate the EV ICD defibrillation testing success rate at implant is greater than an OPC of 88%. H0: p ≤ 0.88 HA: p > 0.88, where p denotes the probability of EV ICD defibrillation success at implant; Test type: Superiority — The pre-specified OPC for the EV ICD defibrillation testing success at implant is 0.88. If the lower confidence bound of two-sided 95% confidence interval for the proportion of EV ICD patients achieving defibrillation testing success at implant exceeds 0.88, the primary efficacy objective will be met. The primary efficacy objective will be evaluated using a one-proportion binomial exact test along with a two-sided 95% Clopper-Pearson confidence bound; p < 0.0001, One-proportion binomial exact test — A priori threshold for statistical significance is 0.025; Proportion = 98.7, 95% CI 2-sided [96.6 to 99.6]

ADVERSE EVENTS:
Time Frame: Pivotal: Among the 356 enrolled subjects, the average follow-up duration from enrollment to last documented contact was 309 days. Forty exited the study without having an implant attempt. Among the 316 subjects who underwent an implant attempt of the EV ICD System, the average follow-up duration from implant attempt to last documented contact was 322 days (range: 10 - 924 days). EV ICD CA: Consent to implant, then 30 days post implant and at 6 month intervals until study closure (10 months).
Description: All adverse events (AEs) are collected throughout the study duration, starting at the time the Informed Consent Form is signed.
  Reporting of these events to Medtronic will occur on an Adverse Event eCRF, including a description of AE, date of onset of AE, date of awareness of site, treatment, resolution, assessment of both the seriousness and the relatedness to the system and/or procedure.
  The Pivotal Study used MedDRA 25.0, the Continued Access Study used MedDRA 26.0
Groups:
- Enrolled Pivotal: Subjects enrolled in the Extravascular ICD Pivotal Study
- Enrolled Continued Access: Subjects enrolled in the Extravascular ICD Continued Access Study (Used MedDRA 26.0)
Arm/Group | Enrolled Pivotal | Enrolled Continued Access
All-Cause Mortality (participants affected / at risk) | 7/356 | 1/37
Serious Adverse Events (participants affected / at risk) | 172/356 | 6/37
Other Adverse Events (participants affected / at risk) | 20/356 | 2/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Pivotal (N=356) | Enrolled Continued Access (N=37)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infection (Cardiac disorders) | 4 (4) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmic Storm (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 14 (16) | 0 (0)
Atrial flutter (Cardiac disorders) | 3 (3) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 15 (18) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 7 (9) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 2 (2) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 3 (3) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
Device inappropriate shock delivery (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 3 (3) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 8 (13) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 9 (10) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Basedow's disease (Endocrine disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 3 (3) | 0 (0)
Implant site haemorrhage (General disorders) | 1 (1) | 0 (0)
Implant site pain (General disorders) | 2 (2) | 0 (0)
Medical device site discomfort (General disorders) | 1 (1) | 0 (0)
Medical device site pain (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Phantom shocks (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 2 (2) | 0 (0)
Eosinophilic granulomatosis with polyangiitis (Immune system disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Chronic hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 2 (2) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Postoperative wound infection (Infections and infestations) | 4 (4) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Spontaneous bacterial peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Systemic infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Device placement issue (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site impaired healing (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nail avulsion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Facial spasm (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Small fibre neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 7 (7) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Device computer issue (Product Issues) | 1 (1) | 0 (0)
Device inappropriate shock delivery (Product Issues) | 23 (29) | 2 (2)
Device inversion (Product Issues) | 4 (4) | 0 (0)
Device lead damage (Product Issues) | 2 (2) | 0 (0)
Lead dislodgement (Product Issues) | 10 (11) | 1 (1)
Oversensing (Product Issues) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Bladder stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Acquired phimosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypopharyngeal synechiae (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 0 (0)
Hypotension (Vascular disorders) | 11 (11) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 1 (2) | 0 (0)
Microangiopathy (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Device pacing issue (Product Issues) | 0 (0) | 1 (1) — Elevated defibrillation thresholds
Emphysematous cystitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Pivotal (N=356) | Enrolled Continued Access (N=37)
Infections and infestations (Infections and infestations) | 20 (20) | 0 (0) — COVID-19
Pain in area of device pocket (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, contracts allow investigators to publish study results per the protocol and publication plan. Investigators and participating institutions will provide any publication of study data generated by the Investigator and/or participating institution to Medtronic for review prior to submission to determine if confidential information ("CI") is included and to check for technical correctness. Medtronic may not censor/interfere with the publication beyond the extent necessary to protect CI.

DOCUMENTS (2):
  • Study Protocol (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/80/NCT04060680/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT04060680/SAP_001.pdf